CLINICAL TRIAL: NCT06354257
Title: A Phase 1, Open-label, Fixed Sequence, 1-way Drug-drug Interaction Study to Investigate the Pharmacokinetics of GSK3036656 and an Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel When the Oral Contraceptive is Administered Alone and in Combination With GSK3036656 in Healthy Female Participants of Nonchildbearing Potential Aged 18-65 Years of Age
Brief Title: A Study to Investigate the Pharmacokinetics of a Combined Oral Contraceptive When Given Alone and in Combination With GSK3036656 in Female Participants of Non-childbearing Potential Aged 18 to 65 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 220104
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis
Keywords: Oral contraceptive; GSK3036656; Fixed sequence; Ethinyl Estradiol; Levonorgestrel; Drug interaction
MeSH Terms: conditions — Tuberculosis | interventions — ethinyl estradiol, levonorgestrel drug combination; GSK656

STUDY DESIGN:
Intervention Model Description: Fixed sequence
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined Participants Group (Experimental): Participants received a dose of Microgynon [0.03 mg Ethinyl Estradiol (EE)/0.15 mg Levonorgestrel (LNG)] on Day 1 of Treatment Period 1. In Treatment Period 2, they received GSK3036656 40 mg on Day 4 followed by GSK3036656 20 mg once daily from Day 5 to Day 14. In Treatment Period 3, participants received Microgynon (EE/LNG) along with GSK3036656 20 mg on Day 15, followed by GSK3036656 20 mg once daily from Day 16 to Day 17.
  Interventions: Drug: Microgynon; Drug: GSK3036656

INTERVENTIONS:
Drug: Microgynon — Participants received 1 dose of Microgynon (0.03 mg EE/0.15 mg LNG) on Day 1 of Treatment Period 1 and 1 dose co-administered with GSK3036656 20 mg on Day 15 of Treatment Period 3.
Drug: GSK3036656 — Participants received 1 loading dose of 40 mg on Day 4 and a dose of 20 mg on Days 5 to 14 once daily in Treatment Period 2. In Treatment Period 3, participants received one 20 mg dose along with Microgynon (0.03 mg EE/0.15 mg LNG) on Day 15 after which a 20 mg dose on Days 17 and 18 once daily.

SUMMARY:
The purpose of this study is to provide data showing if there are any effects of GSK3036656 on a combined oral contraceptive containing Ethinyl Estradiol (EE) and Levonorgestrel (LNG), which will help inform future studies on suitable contraceptive measures to be used.

ELIGIBILITY:
Inclusion Criteria:

Age:

1. Participant was 18 to 65 years of age, inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics:
2. Participants were healthy or compensated, as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
3. Creatinine clearance was >= 75 mL/min.
4. Echocardiogram was normal or showed normal left ventricular function; at most trace to mild valvular regurgitation was allowed, with no valvular stenosis.

   Weight:
5. Body weight was >= 45.0 kg (99 lbs), and body mass index was within the range 18.5 to 31.0 kg/m² (inclusive).

   Sex:
6. Female participants were of Nonchildbearing Potential (WONCBP).

   Women in the following categories were considered WONCBP:

   Permanently sterile due to one of the following procedures:
   1. Documented hysterectomy.
   2. Documented bilateral salpingectomy.
   3. Documented bilateral oophorectomy.

   Postmenopausal females. A postmenopausal state was defined as no menses for 12 months without an alternative medical cause.
   * A high follicle-stimulating hormone (FSH) level in the postmenopausal range could have been used to confirm a postmenopausal state in women not using hormonal contraception or hormone replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with >1 FSH measurement was required within the screening period.
   * Females on HRT and whose menopausal status was in doubt discontinued HRT >= 30 days prior to the start of Treatment Period 1 to allow confirmation of postmenopausal status before study enrolment.

   Informed Consent:
7. Participant was capable of giving signed informed consent, which included compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

Medical History:

1. History of known cardiac valve abnormalities.

   Laboratory Assessments:
2. Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study treatment.
3. Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study treatment, and positive on reflex to hepatitis C RNA.
4. Positive HIV-1 and -2 antigen/antibody immunoassay at Screening.
5. Alanine aminotransferase (ALT) > 1.5×ULN. A single repeat of ALT was allowed within a single screening period to determine eligibility.
6. Bilirubin > 1.5×ULN (isolated bilirubin > 1.5×ULN was acceptable if bilirubin was fractionated and direct bilirubin was < 35%).
7. Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should have precluded participation in the study of an investigational compound.
8. Participants with haemoglobin < 8.0 g/dL.
9. Any Grade 2 to 4 laboratory abnormality at Screening-except creatine phosphokinase, lipid abnormalities, and ALT (as above)-excluded a participant unless the investigator provided a compelling explanation and had sponsor assent. A single repeat of any laboratory abnormality was allowed within a single screening period.
10. Positive test result for drugs of abuse (including marijuana), alcohol, or cotinine at Screening or before the first study dose.

    Prior/Concomitant Therapy:
11. Participants were unable to refrain from using prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's wort), within 7 days prior to the first dose and throughout the study.

    Levothyroxine and omeprazole were allowed if participants had been on a stable dose for >= 1 month prior to Treatment Period 1 and maintained the same dose. Microgynon was administered >= 1 hour after levothyroxine or omeprazole. Other medications were allowed on a case-by-case basis with medical monitor and GSK ganfeborole team approval.
12. Participants received any vaccine within 30 days prior to study treatment.
13. Participants were unwilling to abstain from excessive consumption of caffeine, grapefruit, grapefruit juice, Seville oranges, blood oranges, pomelos, or their juices within 7 days prior to first dose through study end.
14. Participants who had undergone IVF or assisted reproductive techniques within 9 months prior to screening, were currently participating, or planned such procedures during the following year were excluded.

    Prior/Concurrent Clinical Study Experience:
15. Participants had taken part in another clinical study within 30 days, 5 half-lives + 10 days, or 2× duration of the investigational product's biological effect (whichever was longer).
16. Study participation resulted in donation of blood or blood products > 500 mL within 56 days.

    Diagnostic Assessments:
17. Significant arrhythmia or ECG findings, in the opinion of the investigator or GSK Medical Monitor, would have interfered with participant safety.
18. Exclusion criteria for screening ECG:

    Heart rate < 50 or > 100 bpm

    QTcF interval > 450 ms

    Other Exclusion Criteria:
19. Participants with vitiligo.
20. Participants with hypertension or Type 2 diabetes that could not be controlled with diet and exercise alone.
21. History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake > 14 units.
22. Use of tobacco- or nicotine-containing products within 3 months prior to Screening.
23. History of sensitivity to any study medications or components, or any allergy that, in the investigator's or medical monitor's opinion, contraindicated participation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Combined Participants Group includes all participants from the 3 treatment periods combined. This group was used to summarize Participant Flow and Baseline Characteristics in the study.
Period: Treatment Period 1
Arm/Group | Combined Participants Group
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment Period 2
Arm/Group | Combined Participants Group
Started | 19
Completed | 18
Not Completed | 1
Not completed — Adverse Event | 1
Period: Treatment Period 3
Arm/Group | Combined Participants Group
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined Participants Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 53.6 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Drug Concentration (AUC) From Time Zero Extrapolated to Infinity (AUC[0-inf]) After a Single Dose of EE and LNG
Description: AUC(0-inf) is defined as the area under the concentration-time curve from time 0 extrapolated to infinity and was calculated by using a non-compartmental analysis.
Time Frame: At Day 1 for the Treatment Period 1: Microgynon Group and at Day 15 for the Treatment Period 3: Microgynon + GSK3036656 Group
Population: The analysis was performed on the Pharmacokinetic (PK) Set which includes all the participants from the Safety Set (SS) who had at least 1 non-missing PK assessment. This population is defined according to the treatment actually received by the participants and comprises only those with the specified PK parameter available for summary computation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picogram per milliliter (h*pg/mL)
Groups:
- Treatment Period 1: Microgynon Group: Participants received a single dose of Microgynon (0.03 mg EE/0.15 mg LNG) on Day 1 of Treatment Period 1.
- Treatment Period 3: Microgynon + GSK3036656 Group: Participants received Microgynon (EE/LNG) along with GSK3036656 20 mg on Day 15, followed by GSK3036656 20 mg once daily from Day 16 to Day 17 during Treatment Period 3.
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 8 | 9
hour*picogram per milliliter (h*pg/mL)
  EE, Day 1: number analyzed (Participants) | 6 | 0
  EE, Day 1 | 627.11 (53.0) |
  EE, Day 15: number analyzed (Participants) | 0 | 8
  EE, Day 15 |  | 552.01 (51.0)
  LNG, Day 1: number analyzed (Participants) | 8 | 0
  LNG, Day 1 | 24651.76 (113.2) |
  LNG, Day 15: number analyzed (Participants) | 0 | 9
  LNG, Day 15 |  | 30334.48 (94.2)
Statistical Analysis 1: Comparison: Treatment Period 1: Microgynon Group vs Treatment Period 3: Microgynon + GSK3036656 Group; A confirmatory hypothesis testing to test the effect of GSK3036656 on the AUC(0-inf) of EE; Test type: Equivalence — The 90% CI for each ratio was compared to 0.8 and 1.25; Mixed Models Analysis; Analysis was performed using linear mixed effect models with treatment as a fixed effect and subject as a random effect; Geometric mean ratio = 0.88, 90% CI 2-sided [0.55 to 1.41] — One-sided tests (alpha=0.05) were used. 90% CIs for each ratio were compared to 0.8-1.25. No drug interaction is shown if CIs for AUC(0-inf) and Cmax of EE and LNG fall within 0.8-1.25
Statistical Analysis 2: Comparison: Treatment Period 1: Microgynon Group vs Treatment Period 3: Microgynon + GSK3036656 Group; A confirmatory hypothesis testing to test the effect of GSK3036656 on the AUC(0-inf) of LNG; Test type: Equivalence — The 90% CI for each ratio was compared to 0.8 and 1.25; Mixed Models Analysis; Analysis was performed using linear mixed effect models with treatment as a fixed effect and subject as a random effect; Geometric mean ratio = 1.10, 90% CI 2-sided [0.98 to 1.23] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) After a Single Dose of EE and LNG
Description: Cmax is defined as the maximum observed plasma concentration determined directly from the concentration-time data and was calculated by using a non-compartmental analysis.
Time Frame: as for outcome 1
Population: The analysis was performed on the PK Set which includes all the participants from the SS who had at least 1 non-missing PK assessment. This population is defined according to the treatment actually received by the participants and comprises only those with the specified PK parameter available for summary computation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 19 | 18
picogram per milliliter (pg/mL)
  EE, Day 1: number analyzed (Participants) | 19 | 0
  EE, Day 1 | 50.86 (32.7) |
  EE, Day 15: number analyzed (Participants) | 0 | 18
  EE, Day 15 |  | 48.96 (24.5)
  LNG, Day 1: number analyzed (Participants) | 19 | 0
  LNG, Day 1 | 2599.85 (46.8) |
  LNG, Day 15: number analyzed (Participants) | 0 | 18
  LNG, Day 15 |  | 2828.17 (45.3)
Statistical Analysis 1: Comparison: Treatment Period 1: Microgynon Group vs Treatment Period 3: Microgynon + GSK3036656 Group; A confirmatory hypothesis testing to test the effect of GSK3036656 on the Cmax of EE; Test type: Equivalence — The 90% CI for each ratio was compared to 0.8 and 1.25; Mixed Models Analysis; Analysis was performed using linear mixed effect models with treatment as a fixed effect and subject as a random effect; Geometric mean ratio = 0.96, 90% CI 2-sided [0.85 to 1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment Period 1: Microgynon Group vs Treatment Period 3: Microgynon + GSK3036656 Group; A confirmatory hypothesis testing to test the effect of GSK3036656 on the Cmax of LNG; Test type: Equivalence — The 90% CI for each ratio was compared to 0.8 and 1.25; Mixed Models Analysis; Analysis was performed using linear mixed effect models with treatment as a fixed effect and subject as a random effect; Geometric mean ratio = 1.08, 90% CI 2-sided [0.97 to 1.19] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC Versus Time Curve From Time Zero During a Dosage Interval of Time at Steady State [AUC(0-tau)] of GSK3036656 With EE/LNG
Description: AUC(0-tau) is defined as the area under the concentration-time curve over a dosing interval and was calculated by using a non-compartmental analysis.
Time Frame: At Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 18
hour*nanogram per milliliter (h*ng/mL) | 8372.42 (18.8)

4. Secondary Outcome: Cmax at Steady State of GSK3036656 With EE/LNG
Description: as for outcome 2
Time Frame: At Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 18
nanogram per milliliter (ng/mL) | 600.62 (14.2)

5. Secondary Outcome: Trough Plasma Concentration (Ctau) at Steady State of GSK3036656 With EE/LNG and GSK3036656 Alone
Description: Ctau is defined as the concentration reached by the drug immediately before the next dose is administered.
Time Frame: At Day 8, 10, 12, 15 and 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment Period 2: GSK3036656 Group: Participants received GSK3036656 40 mg on Day 4, followed by GSK3036656 20 mg once daily from Day 5 to Day 14 during Treatment Period 2.
Arm/Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 19 | 18
ng/mL
  Day 8: number analyzed (Participants) | 19 | 0
  Day 8 | 226.92 (17.9) |
  Day 10: number analyzed (Participants) | 19 | 0
  Day 10 | 235.54 (27.5) |
  Day 12: number analyzed (Participants) | 19 | 0
  Day 12 | 243.40 (21.9) |
  Day 15: number analyzed (Participants) | 0 | 18
  Day 15 |  | 251.26 (40.3)
  Day 16: number analyzed (Participants) | 0 | 18
  Day 16 |  | 254.91 (23.0)

6. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) at Steady State of GSK3036656 With EE/LNG
Description: Tmax is defined as a measure of the time required to reach the maximum concentration of the drug, determined directly from the concentration-time data.
Time Frame: At Day 15
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 18
hour | 0.95 [0.4 to 3.0]

7. Secondary Outcome: AUC Versus Time Curve (AUC[0-t]) of EE and LNG Alone and With GSK3036656
Description: AUC(0-t) is defined as area under the plasma drug concentration versus time curve from time zero (pre-dose) to last time of quantifiable concentration and was calculated by using a non-compartmental analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 19 | 18
h*pg/mL
  EE, Day 1: number analyzed (Participants) | 19 | 0
  EE, Day 1 | 447.10 (58.7) |
  EE, Day 15: number analyzed (Participants) | 0 | 18
  EE, Day 15 |  | 363.00 (43.4)
  LNG, Day 1: number analyzed (Participants) | 19 | 0
  LNG, Day 1 | 21182.61 (84.3) |
  LNG, Day 15: number analyzed (Participants) | 0 | 18
  LNG, Day 15 |  | 23287.77 (91.3)

8. Secondary Outcome: Tmax of EE and LNG Alone and With GSK3036656
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 19 | 18
hour
  EE, Day 1: number analyzed (Participants) | 19 | 0
  EE, Day 1 | 0.967 [0.47 to 2.97] |
  EE, Day 15: number analyzed (Participants) | 0 | 18
  EE, Day 15 |  | 1.433 [0.45 to 3.05]
  LNG, Day 1: number analyzed (Participants) | 19 | 0
  LNG, Day 1 | 0.967 [0.92 to 1.93] |
  LNG, Day 15: number analyzed (Participants) | 0 | 18
  LNG, Day 15 |  | 0.967 [0.45 to 2.07]

9. Secondary Outcome: Apparent Terminal Half-life (t1/2) of EE and LNG Alone and With GSK3036656
Description: t1/2 is defined as the time required by the plasma concentration to decline by 50% and was calculated by using a non-compartmental analysis.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 13 | 13
hour
  EE, Day 1: number analyzed (Participants) | 13 | 0
  EE, Day 1 | 19.180 [4.38 to 49.03] |
  EE, Day 15: number analyzed (Participants) | 0 | 10
  EE, Day 15 |  | 10.867 [3.14 to 29.39]
  LNG, Day 1: number analyzed (Participants) | 12 | 0
  LNG, Day 1 | 41.315 [4.00 to 100.00] |
  LNG, Day 15: number analyzed (Participants) | 0 | 13
  LNG, Day 15 |  | 34.697 [4.17 to 118.18]

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is defined as any untoward medical occurrence that, at any dose: resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: From the signing of the informed consent form (a period starting up to 14 days before the first dose on Day 1) up to Day 18
Population: The analysis was performed on the SS which included all the participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Grade 3 or Higher Severity Adverse Events (AEs)
Description: The intensity of AEs was assessed using the Division of Acquired Immunodeficiency Syndrome (DAIDS) criteria Version 2.1 where grades are defined based on numeric criteria as follows Grade 3: severe or medically significant; Grade 4: potentially life-threatening; Grade 5: death. A higher grade indicates greater severity.
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Drug-related AEs Following Administration of Microgynon and Following the Administration of GSK3036656
Description: The drug-related AEs were assessed by the investigator to be possibly, probably or definitely related to the study interventions.
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Withdrawn From the Treatment Due to AEs
Description: Adverse events resulting in withholding of study intervention administration were included in this outcome measure.
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants | 0 | 1 | 0

14. Secondary Outcome: Number of Participants Withdrawn From the Study Due to AEs
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants | 0 | 1 | 0

15. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Importance (PCI)
Description: PCI ECG values are defined as any ECG findings which, in the opinion of the investigator or medical monitor would interfere with the safety of the individual participant. The ECG measurements analyzed are PR Interval, QRS Duration, and QTcF Interval. A value was reported as "high" for a period if it shifted from "low" or "within range" (W/in) at the start of the treatment period but was "high" during or at the end of the same treatment period. A value was reported as "low" for a period if it shifted from "high" or "W/in" at the start of the treatment period but was "low" during or at the end of the same treatment period. A value was reported as "No Change" if it remained unchanged (e.g. High to High), or as "To W/in Range" if it was within range.
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants
  PR Interval, To Low | 0 | 0 | 0
  PR Interval, To W/in Range or No Change | 20 | 19 | 18
  PR Interval, To High | 0 | 0 | 0
  QRS Duration, To Low | 3 | 1 | 3
  QRS Duration, To W/in Range or No Change | 17 | 18 | 15
  QRS Duration, To High | 0 | 0 | 0
  QTcF Interval, To Low | 0 | 0 | 0
  QTcF Interval, To W/in Range or No Change | 20 | 19 | 18
  QTcF Interval, To High | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinical Chemistry Laboratory Values of PCI
Description: The chemistry parameters analyzed are homocysteine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), direct bilirubin, bilirubin, calcium, creatine kinase, potassium, protein, sodium, urea, and glucose. A value was reported as "high" for a period if it shifted from "low" or "within range" (W/in) at the start of the treatment period but was "high" during or at the end of the same treatment period. A value was reported as "low" for a period if it shifted from "high" or "W/in" at the start of the treatment period but was "low" during or at the end of the same treatment period. A value was reported as "No Change" if it remained unchanged (e.g. High to High), or as "To W/in Range" if it was within range.
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Homocysteine, To Low | 0 | 0 | 0
  Homocysteine, To W/in Range or No Change | 19 | 19 | 15
  Homocysteine, To High | 1 | 0 | 3
  ALT, To Low | 0 | 0 | 0
  ALT, To W/in Range or No Change | 20 | 19 | 18
  ALT, To High | 0 | 0 | 0
  AST, To Low: number analyzed (Participants) | 20 | 16 | 15
  AST, To Low | 0 | 0 | 0
  AST, To W/in Range or No Change: number analyzed (Participants) | 20 | 16 | 15
  AST, To W/in Range or No Change | 20 | 16 | 15
  AST, To High: number analyzed (Participants) | 20 | 16 | 15
  AST, To High | 0 | 0 | 0
  Direct Bilirubin, To Low: number analyzed (Participants) | 20 | 18 | 17
  Direct Bilirubin, To Low | 0 | 0 | 0
  Direct Bilirubin, To W/in Range or No Change: number analyzed (Participants) | 20 | 18 | 17
  Direct Bilirubin, To W/in Range or No Change | 20 | 17 | 17
  Direct Bilirubin, To High: number analyzed (Participants) | 20 | 18 | 17
  Direct Bilirubin, To High | 0 | 1 | 0
  Bilirubin, To Low: number analyzed (Participants) | 20 | 18 | 17
  Bilirubin, To Low | 0 | 0 | 0
  Bilirubin, To W/in Range or No Change: number analyzed (Participants) | 20 | 18 | 17
  Bilirubin, To W/in Range or No Change | 20 | 18 | 17
  Bilirubin, To High: number analyzed (Participants) | 20 | 18 | 17
  Bilirubin, To High | 0 | 0 | 0
  Calcium, To Low | 0 | 0 | 0
  Calcium, To W/in Range or No Change | 20 | 19 | 18
  Calcium, To High | 0 | 0 | 0
  Creatine Kinase, To Low | 0 | 0 | 0
  Creatine Kinase, To W/in Range or No Change | 20 | 18 | 18
  Creatine Kinase, To High | 0 | 1 | 0
  Potassium, To Low: number analyzed (Participants) | 20 | 16 | 15
  Potassium, To Low | 0 | 0 | 0
  Potassium, To W/in Range or No Change: number analyzed (Participants) | 20 | 16 | 15
  Potassium, To W/in Range or No Change | 20 | 16 | 15
  Potassium, To High: number analyzed (Participants) | 20 | 16 | 15
  Potassium, To High | 0 | 0 | 0
  Protein, To Low | 0 | 0 | 0
  Protein, To W/in Range or No Change | 20 | 19 | 18
  Protein, To High | 0 | 0 | 0
  Sodium, To Low | 0 | 0 | 0
  Sodium, To W/in Range or No Change | 20 | 19 | 18
  Sodium, To High | 0 | 0 | 0
  Urea, To Low | 0 | 0 | 0
  Urea, To W/in Range or No Change | 19 | 19 | 18
  Urea, To High | 1 | 0 | 0
  Glucose, To Low: number analyzed (Participants) | 19 | 18 | 18
  Glucose, To Low | 0 | 0 | 0
  Glucose, To W/in Range or No Change: number analyzed (Participants) | 19 | 18 | 18
  Glucose, To W/in Range or No Change | 19 | 18 | 18
  Glucose, To High: number analyzed (Participants) | 19 | 18 | 18
  Glucose, To High | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Haematology Laboratory Values of PCI
Description: The analyzed hematology parameters are reticulocytes/erythrocytes, monocytes/leukocytes, erythrocytes, basophils/leukocytes, eosinophils/leukocytes, mean corpuscular hemoglobin, hematocrit, hemoglobin, lymphocytes, neutrophils, and platelets. A value was reported as "high" for a period if it shifted from "low" or "within range" (W/in) at the start of the treatment period but was "high" during or at the end of the same treatment period. A value was reported as "low" for a period if it shifted from "high" or "W/in" at the start of the treatment period but was "low" during or at the end of the same treatment period. A value was reported as "No Change" if it remained unchanged (e.g. High to High), or as "To W/in Range" if it was within range.
Time Frame: From Day 1 up to Day 18
Population: The analysis was performed on the SS which included all the participants who received at least one dose of study medication. Only participants for whom haematology data were available were included in the analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 18 | 17
Participants
  Basophils/Leukocytes, To Low | 7 | 1 | 1
  Basophils/Leukocytes, To W/in Range or No Change | 13 | 17 | 16
  Basophils/Leukocytes, To High | 0 | 0 | 0
  Eosinophils/Leukocytes, To Low | 1 | 0 | 2
  Eosinophils/Leukocytes, To W/in Range or No Change | 19 | 14 | 15
  Eosinophils/Leukocytes, To High | 0 | 4 | 0
  Monocytes/Leukocytes, To Low | 0 | 0 | 0
  Monocytes/Leukocytes, To W/in Range or No Change | 20 | 17 | 17
  Monocytes/Leukocytes, To High | 0 | 1 | 0
  Erythrocytes, To Low | 0 | 5 | 0
  Erythrocytes, To W/in Range or No Change | 20 | 13 | 17
  Erythrocytes, To High | 0 | 0 | 0
  Reticulocytes/Erythrocytes, To Low | 0 | 0 | 0
  Reticulocytes/Erythrocytes, To W/in Range or No Change | 19 | 16 | 16
  Reticulocytes/Erythrocytes, To High | 1 | 2 | 1
  Mean Corpuscular Hemoglobin, To Low | 0 | 0 | 0
  Mean Corpuscular Hemoglobin, To W/in Range or No Change | 20 | 18 | 17
  Mean Corpuscular Hemoglobin, To High | 0 | 0 | 0
  Hematocrit, To Low | 0 | 0 | 0
  Hematocrit, To W/in Range or No Change | 20 | 18 | 17
  Hematocrit, To High | 0 | 0 | 0
  Hemoglobin, To Low | 0 | 0 | 0
  Hemoglobin, To W/in Range or No Change | 20 | 18 | 17
  Hemoglobin, To High | 0 | 0 | 0
  Lymphocytes, To Low | 0 | 0 | 0
  Lymphocytes, To W/in Range or No Change | 20 | 18 | 17
  Lymphocytes, To High | 0 | 0 | 0
  Neutrophils, To Low | 0 | 0 | 0
  Neutrophils, To W/in Range or No Change | 20 | 18 | 17
  Neutrophils, To High | 0 | 0 | 0
  Platelets, To Low | 0 | 0 | 0
  Platelets, To W/in Range or No Change | 20 | 18 | 17
  Platelets, To High | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Vital Signs Parameters of PCI
Description: The analyzed vital signs are systolic blood pressure, diastolic blood pressure, heart rate, body temperature, and respiration rate. A value was reported as "high" for a period if it shifted from "low" or "within range" (W/in) at the start of the treatment period but was "high" during or at the end of the same treatment period. A value was reported as "low" for a period if it shifted from "high" or "W/in" at the start of the treatment period but was "low" during or at the end of the same treatment period. A value was reported as "No Change" if it remained unchanged (e.g. High to High), or as "To W/in Range" if it was within range.
Time Frame: From Day 1 up to Day 18
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Diastolic Blood Pressure, To Low | 0 | 0 | 0
  Diastolic Blood Pressure, To w/in Range or No Change | 20 | 19 | 18
  Diastolic Blood Pressure, To High | 0 | 0 | 0
  Pulse Rate, To Low | 0 | 0 | 0
  Pulse Rate, To w/in Range or No Change | 20 | 19 | 18
  Pulse Rate, To High | 0 | 0 | 0
  Respiratory Rate, To Low | 0 | 0 | 0
  Respiratory Rate, To w/in Range or No Change | 20 | 19 | 18
  Respiratory Rate, To High | 0 | 0 | 0
  Systolic Blood Pressure, To Low | 0 | 0 | 0
  Systolic Blood Pressure, To w/in Range or No Change | 20 | 19 | 18
  Systolic Blood Pressure, To High | 0 | 0 | 0
  Temperature, To Low | 0 | 0 | 0
  Temperature, To w/in Range or No Change | 20 | 19 | 18
  Temperature, To High | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from Day 1 (first study dose) up to Day 18. Serious Adverse Events were reported from the signing of the informed consent form (a period starting up to 14 days before the first dose on Day 1) up to Day 18
Arm/Group | Treatment Period 1: Microgynon Group | Treatment Period 2: GSK3036656 Group | Treatment Period 3: Microgynon + GSK3036656 Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 4/20 | 1/19 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1: Microgynon Group (N=20) | Treatment Period 2: GSK3036656 Group (N=19) | Treatment Period 3: Microgynon + GSK3036656 Group (N=18)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT06354257/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT06354257/SAP_001.pdf